CLINICAL TRIAL: NCT05458128
Title: An Open-Label Study to Evaluate the Long-Term Safety and Effectiveness of Pitolisant in Adult Patients With Idiopathic Hypersomnia Who Completed Study HBS-101-CL-010
Brief Title: A Long-Term Safety and Effectiveness Study to Evaluate Pitolisant in Adult Patients With Idiopathic Hypersomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harmony Biosciences Management, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBS-101-CL-011
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Idiopathic Hypersomnia; Excessive Daytime Sleepiness
Keywords: pitolisant; histamine; sleepiness; IH
MeSH Terms: conditions — Idiopathic Hypersomnia; Disorders of Excessive Somnolence; Sleepiness | interventions — pitolisant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pitolisant (Other): Week 1: 8.9 mg pitolisant administered once daily in the morning upon wakening; Week 2: 17.8 mg pitolisant administered once daily in the morning upon wakening; Weeks 3 through end of treatment: 17.8 mg to 35.6 mg pitolisant administered once daily in the morning upon wakening.
  Interventions: Drug: Pitolisant

INTERVENTIONS:
Drug: Pitolisant — Pitolisant 4.45 mg tablets
  Pitolisant 17.8 mg tablets

SUMMARY:
The primary objective of this study is to assess the long-term safety and effectiveness of pitolisant in patients with idiopathic hypersomnia (IH) who completed the Double-Blind Randomized Withdrawal Phase of study HBS-101-CL-010.

DETAILED DESCRIPTION:
This is a Phase 3 open-label study to evaluate the long-term safety and effectiveness of pitolisant in adult patients with IH. Patients who complete the Double-Blind Randomized Withdrawal Phase of study HBS-101-CL-010 (i.e., completed the End-of-Treatment [EOT] Visit/Visit 5 in the HBS-101-CL-010 study) and who continue to meet eligibility criteria for study HBS-101-CL-011 are eligible for enrollment.

Enrolled patients will be dispensed open-label pitolisant and may be titrated up to a maximum dose of 35.6 mg, based on the Investigator's assessment of safety/tolerability and effectiveness, during a 3-week Titration Period (Day 1 to Day 21) in accordance with the schedule:

* Week 1 (Day 1-7), 8.9 mg
* Week 2 (Day 8-14), 17.8 mg
* Week 3 (Day 15-21), 35.6 mg

The Long-Term Dosing Period will begin on Day 22 and will continue until the patient discontinues from the study or the Sponsor elects to terminate the study (i.e., End-of-Study [EOS]).

An on-site study visit will occur approximately 180 days after Visit 2 on Day 202 (Visit 3). On-site study visits will occur approximately every 6 months and telephone contacts (TCs) approximately every one month in between until the patient withdraws from the study or the study is terminated by the Sponsor. The dose of pitolisant may be adjusted (higher or lower) in increments of 4.45 mg starting at 8.9 mg up to 35.6 mg during the Long-Term Dosing Period based on Investigator assessment of safety/tolerability and effectiveness.

All patients will receive safety follow-up TCs from the study site 15 days and 30 days after their final dose of pitolisant, to assess for adverse events (AEs) and concomitant medication use.

ELIGIBILITY:
Inclusion Criteria:

1. Is able to provide voluntary, informed consent.
2. Completed the Double-Blind Randomized Withdrawal Phase (EOT/Visit 5) from the HBS-101-CL-010 study.
3. A patient who is a female of child-bearing potential must have a negative urine pregnancy test at the Screening Visit. A patient who is a female of child-bearing potential must agree to remain abstinent or use an effective method of non-hormonal contraception to prevent pregnancy for the duration of the study and for 21 days after final dose of study drug.
4. Must have a negative result on urine drug screen at the Screening Visit, except for medications that are prescribed by a healthcare provider for medical conditions.
5. In the opinion of the Investigator, the patient is capable of understanding and complying with the protocol and administration of oral study drug.

Exclusion Criteria:

1. Does not agree to discontinue any prohibited medication or substances listed in the protocol.
2. Is currently breastfeeding or planning to breastfeed over the course of the study. Lactating women must agree not to breastfeed for the duration of the study and for 21 days after final dose of study drug.
3. Participation in an interventional research study with an investigational medication or device, other than pitolisant, for the duration of the study.
4. Has a diagnosis of end-stage renal disease (ESRD; estimated glomerular filtration rate [eGFR] of <15 mL/minute/1.73 m2) or severe hepatic impairment (Child-Pugh C).
5. Is receiving or is unable to discontinue a medication known to prolong the QT interval.
6. Has a significant risk of committing suicide or suicidality based on history; routine psychiatric examination; Investigator's judgment; or who has an answer of "yes" on any question other than questions 1 to 3 or "yes" on any question in the suicidal behavior section of the C-SSRS, Since Last Visit.
7. Based on the judgment of the Investigator, is unsuitable for the study for any reason, including but not limited to an unstable or uncontrolled medical condition or one that might interfere with the conduct of the study, confound interpretation of study results, pose a health risk to the patient, or compromise the integrity of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of pitolisant | Up to approximately 3 years
  Incidence of adverse events (AEs)
Excessive daytime sleepiness | Up to approximately 3 years
  Change from Baseline in Epworth Sleepiness Scale (ESS) score
  The score of the Epworth Sleepiness Scale ranges from 0 to 24. A decrease in score represents an improvement in excessive daytime sleepiness.

SECONDARY OUTCOMES:
Symptoms of idiopathic hypersomnia | Up to approximately 3 years
  Change from Baseline in Idiopathic Hypersomnia Severity Scale (IHSS)
  The score of the IHSS ranges from 0 to 50. A decrease in score represents an improvement in symptoms of idiopathic hypersomnia.
Symptoms of idiopathic hypersomnia | Up to approximately 3 years
  Change from Baseline in Clinical Global Impression of Severity (CGI-S) for IH
  The CGI-S is a five-item scale that ranges from none to very severe. An assessment of less severe symptoms represents an improvement in the clinician's perception of the patient's overall clinical status related to idiopathic hypersomnia.
Symptoms of idiopathic hypersomnia | Up to approximately 3 years
  Change from Baseline in Patient Global Impression of Severity (PGI-S) for EDS
  The PGI-S is a five-item scale that ranges from none to very severe. An assessment of less severe symptoms represents an improvement in the patient's perception of the severity of their excessive daytime sleepiness.
Functional outcomes of sleep | Up to approximately 3 years
  Change from Baseline in Functional Outcomes of Sleep Questionnaire 10-item version (FOSQ-10)
  The score of the FOSQ-10 ranges from 5 to 20. An increase in score represents an improvement in the patient's impression of the impact of hypersomnia on multiple activities of everyday living.
Sleep related impairments during wakefulness | Up to approximately 3 years
  Change from Baseline in Patient-Reported Outcomes Measurement Information System Sleep-Related Impairment Item Bank v1.0-Short Form 8a (PROMIS-SRI 8a)
  The score of the PROMIS-SRI 8a ranges from 8-40. A decrease in score represents an improvement in the patient's impression of the impact of hypersomnia on multiple activities of everyday living.
Sleep inertia | Up to approximately 3 years
  Change from Baseline in Sleep Inertia Questionnaire (SIQ)
  The SIQ ranges from 21 to 105. A decrease in score represents an improvement in the patient's ability to wake up after sleep.

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Cedars-Sinai Medical Towers, Los Angeles, California
  - Sleep Medicine Specialists of California, San Ramon, California
  - Meris Clinical Research, Brandon, Florida
  - St. Francis Medical Institute, Clearwater, Florida
  - Florida Pediatric Research Institute, Winter Park, Florida
  - Neurotrials Research Inc., Atlanta, Georgia
  - NorthShore University Health System, Glenview, Illinois
  - OSF HealthCare Saint Francis Medical Center, Peoria, Illinois
  - Western Michigan University Homer Stryker MD School of Medicine, Kalamazoo, Michigan
  - Clinical Neurophysiology Services, Sterling Heights, Michigan
  - St. Luke's Sleep Medicine and Research Center, Chesterfield, Missouri
  - Clayton Sleep Institute, St Louis, Missouri
  - Great Plains Health, North Platte, Nebraska
  - Sleep Dynamics, Neptune City, New Jersey
  - Northwell Health, New Hyde Park, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - ARSM Research, Huntersville, North Carolina
  - NeuroScience Research Center, LLC, Canton, Ohio
  - Intrepid Research, LLC, Cincinnati, Ohio
  - Ohio Sleep Medicine and Neuroscience Institue, Dublin, Ohio
  - North Star Medical Research, Middleburg, Ohio
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Respiratory Specialists, Wyomissing, Pennsylvania
  - Bogan Sleep Consultants, Columbia, South Carolina
  - Lowcountry Lung Critical Care, North Charleston, South Carolina
  - Neurology Clinic, P.C., Cordova, Tennessee
  - FutureSearch Trials of Neurology LP, Austin, Texas
  - Central Texas Neurology Consultants, PA, Round Rock, Texas
  - Comprehensive Sleep Medicine Associates, Sugar Land, Texas
  - Northwest Houston Neurology and Sleep, Tomball, Texas
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No